CLINICAL TRIAL: NCT04712942
Title: Treatment of MDS/AML Patients With an Impending Hematological Relapse With Azacitidine Alone or in Combination With PEvonedistat - a Randomized Phase 2 Trial
Brief Title: Treatment of MDS/AML Patients With an Impending Hematological Relapse With AZA or ATA and Pevonedistat
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Uwe Platzbecker, Prof. Dr., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHAPE
Record Dates: First submitted 2020-12-18; First posted 2021-01-19 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Acute Myeloid Leukemia in Remission; Myelodysplastic Syndromes; Minimal Residual Disease
MeSH Terms: conditions — Myelodysplastic Syndromes; Neoplasm, Residual | interventions — pevonedistat; Azacitidine

STUDY DESIGN:
Intervention Model Description: With Cross-Over option
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pevonedistat + azacitidine (Experimental): pevonedistat in combination with azacitidine
  Interventions: Drug: Pevonedistat; Drug: Azacitidine
- azacitidine monotherapy (Other): administration of azacitidine monotherapy
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Pevonedistat — Patients receive pevonedistat at 20 mg/m2 i.v. (d1,3,5, q4w) up to 12 cycles
  Arms: pevonedistat + azacitidine
Drug: Azacitidine — azacitidine is given at a standard dose of 75 mg/m² (d1-7 or 1-5,8,9, q4w) up to 12 cycles

SUMMARY:
MDS/AML with MRD and impending relapse after allogeneic stem cell transplantation and/or conventional chemotherapy

DETAILED DESCRIPTION:
Experimental arm: pevonedistat in combination with azacitidine Control arm: azacitidine alone

With the following modifications:

* Patients on the azacitidine arm and still MRD+ at 3 months but without hematological relapse can cross over to the combination arm
* Cross over into the combination arm is possible any time up to 9 months of study treatment if initially responding patients (at 3 months) on AZA monotherapy become MRD positive again
* Maximum treatment duration of 1 year
* Patients receive pevonedistat at 20 mg/m2 i.v. (d1,3,5, q4w); azacitidine is given at a standard dose of 75 mg/m² i.v. or s.c. (d1-7 or 1-5,8,9, q4w)

ELIGIBILITY:
Inclusion Criteria:

* AML or MDS
* continuing first CR after conventional intensive chemotherapy OR continuing CR after alloSCT
* Confirmed MRD positivity (assessed by central lab) as defined by:

  * NPM1mut status >1% in peripheral blood or bone marrow in NPM1 mutated patients at diagnosis or
  * Patients after allogeneic transplantation, who were NPM1 unmutated at diagnosis and have a blood or marrow CD34/CD117 chimerism <80%

Exclusion Criteria:

Compliance with major study procedures

* Patient does not accept bone marrow sampling during screening, primary end point visit and after the treatment.
* Patient does not accept several blood sampling during screening, treatment (up to bi-daily) and after the treatment.

Safety

* Inadequate organ function as defined in the list below:

  * White blood cell (WBC) count > 50 Gpt/L before administration of pevonedistat on Cycle 1 Day 1
  * Absolute neutrophil count (ANC) < 1.5 Gpt/L
  * Platelets < 100 Gpt/L
  * Albumin < 2.7 g/dL
  * Creatinine clearance < 30 mL/min (Cockcroft und Gault formula)
  * Total bilirubin > 1.5xupper limit of normal (ULN) except in patients with Gilbert's syndrome. Patients with Gilbert's syndrome may be enrolled if direct bilirubin > 1.5x ULN of the direct bilirubin.
  * Both Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 3.0 ULN
* ECOG performance status of ≥2

Concomitant Diseases

* Hematological relapse
* Liver cirrhosis or severe pre-existing hepatic impairment
* Known severe cardiopulmonary disease (e.g. unstable angina, congestive heart failure NYHA III or IV, myocardial infarction within 6 months prior to screening, symptomatic cardiomyopathy, clinically significant arrhythmia, clinically significant pulmonary hypertension requiring pharmacologic therapy)
* Uncontrolled high blood pressure (i.e. systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg)
* Confirmed prolonged rate corrected QT interval ≥ 500 msec, calculated according to institutional guidelines (Screening ECG)
* Confirmed left ventricular ejection fraction < 50% as assessed by echocardiogram or radionuclide angiography (Screening TTE)
* Known moderate to severe symptomatic chronic obstructive pulmonary disease, interstitial lung disease, or pulmonary fibrosis
* Active uncontrolled infection or severe infectious disease, such as severe pneumonia, meningitis, or septicemia
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Known Human Immunodeficiency Virus (HIV 1/2 antibodies)
* Known active Hepatitis B (i.e. HBsAg reactive) or Hepatitis C (i.e., HCV RNA [qualitative] is detected). NOTE: Patients who have isolated positive hepatitis B core antibody (i.e. in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load.
* Major surgery within 14 days of randomization or a scheduled surgery during study period
* Known central nervous system (CNS) involvement
* Diagnosis or treatment for another malignancy within 2 years before randomization. (NOTE: Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone resection. Prior diagnosis of myelodysplasia, myeloproliferative neoplasm, or aplastic anemia and treatment for that diagnosis does not lead to exclusion)
* Any evidence of residual disease of another malignancy
* Patients with uncontrolled coagulopathy or bleeding disorder
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Unexpected effect of HMA monotherapy

* Prior HMA failure
* Prior HMA treatment without subsequent allogeneic transplantation

Interfering Treatments

* Any ongoing therapy with investigational agents or chemotherapeutic agents active against MDS or AML
* BCRP inhibitors (for exceptions, see section 5.7.5) are not permitted during the study and should be stopped 14 days before first dose of the study drug

Exclusion criteria regarding special restrictions for females of childbearing potential

* Current or planned pregnancy or nursing women (negative urine or serum pregnancy test within 3 days prior to receiving study treatment is needed. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test needs to be required.)
* Female patients of childbearing potential, who are not using or not willing to use 1 highly effective method and 1 additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s).

Exclusion criteria regarding special restrictions for males, even if surgically sterilized (i.e. status post vasectomy)

* Male patients, who do not agree to use an adequate method of contraception, starting with the first dose of study therapy during the entire study treatment period and through 4 months after the last dose of study drug. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s).

Regulatory requirements

* Age under 18 years at registration
* Inability to provide written informed consent
* Subject without legal capacity who is unable to understand the nature, scope, significance and consequences of this clinical trial
* Simultaneous participation in another interventional clinical trial or participation in any clinical trial involving administration of an investigational medicinal product within 30 days prior to SHAPE trial beginning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Measurable residual disease (MRD) status after 3 months of treatment | 3 months after start of treatment
  To show that pevonedistat and azacitidine are more effective compared to azacitidine alone with regard to achievement of MRD negativity after 3 months of treatment.
  MRD assessment is carried out as determination of the NPM1mut status or as CD34/CD117 chimerism analysis.

SECONDARY OUTCOMES:
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 25 months
  To describe and compare outcome measures between two strategies: pevonedistat and azacitidine in combination versus azacitidine alone with cross over option.
Relapse Free Survival | Time from randomization until hematological relapse or death from any cause (whichever comes first), assessed up to 25 Months.
  To describe and compare outcome measures between two strategies: pevonedistat and azacitidine in combination versus azacitidine alone with cross over option.
Impact of treatment assessed by using the validated questionnaires EORTC QLQ-C30. | Time from randomization until hematological relapse or death from any cause (whichever comes first)
  To describe and compare outcome measures between two strategies: pevonedistat and azacitidine in combination versus azacitidine alone with cross over option.
Impact of treatment assessed by using the validated questionnaires EQ-5D-5L. | Time from randomization until hematological relapse or death from any cause (whichever comes first), assessed up to 25 months.
  To describe and compare outcome measures between two strategies: pevonedistat and azacitidine in combination versus azacitidine alone with cross over option.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, Prof. Dr., Principal Investigator — University Leipzig
Locations (14):
- Germany (14):
  - Medizinische Klinik IV - Hämatologie und Onkologie, Universitätsklinikum Aachen, Aachen
  - Zentrum Hämatologie, Onkologie, Palliativmedizin, Helios Klinikum Berlin-Buch GmbH, Berlin
  - Klinik für Innere Medizin III, Hämatologie, Onkologie, Stammzelltransplantation, Klinikum Chemnitz gGmbH, Chemnitz
  - Hämatologie/Internistische Onkologie, Onkologische Tagesklinik, Cottbus
  - Medizinischen Klinik und Poliklinik I / Hämatologie, Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Klinik für Hämatologie, Universitätsklinikum Essen, Essen
  - Universitätsklinik und Poliklinik für Innere Medizin IV, Onkologie, Hämatologie, Universitätsklinikum Halle (Saale), Halle
  - Klinik und Poliklinik für Innere Medizin II/Hämat. - Onkologie, Universitätsklinikum Jena, Jena
  - Klinik für Innere Medizin II/ Hämatologie und Onkologie, Univ.Klinikum Schleswig-Holstein/Campus Kiel, Kiel
  - Medizinische Klinik und Poliklinik I - Hämatologie und Zelltherapie, Hämostaseologie, Leipzig University, Leipzig
  - Innere Medizin A/Hämatologie-Onkologie, Universitätsklinik Münster, Münster
  - Klinik Innere Medizin III - Onko-, Häma- u. Palliativmedizin, Diakonie-Klinikum Schwäbisch Hall gGmbH, Schwäbisch Hall
  - Klinik für Hämatologie, Onkologie & Stammzelltherapie, Helios-Klinikum Schwerin, Schwerin
  - Abteilung für Hämatologie, Onkologie und Palliativmedizin, Robert-Bosch-Krankenhaus Stuttgart, Stuttgart

IPD SHARING:
Plan to Share IPD: No